CLINICAL TRIAL: NCT04705311
Title: The Effect of Pain Neuroscience Education on Patients With Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, Principal Investigator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-1040781-A-N-012021010HR
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Rotator Cuff Injuries; Kinesiophobia; Pain, Postoperative
MeSH Terms: conditions — Rotator Cuff Injuries; Kinesiophobia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pain neuroscience education plus rotator cuff repair rehabilitation (Experimental)
  Interventions: Other: Pain neuroscience education; Behavioral: Rotator cuff repair rehabilitation
- rotator cuff repair rehabilitation (Active Comparator)
  Interventions: Behavioral: Rotator cuff repair rehabilitation

INTERVENTIONS:
Other: Pain neuroscience education — Neurophysiological education of pain allows patients to explore a wider contribution to pain through the knowledge that pain is often an unreliable indicator of the extent or extent of tissue damage. This aims at reconceptualization from biomedical or structural models to actual biological psychosocial pain models.
  Arms: pain neuroscience education plus rotator cuff repair rehabilitation
Behavioral: Rotator cuff repair rehabilitation — Postoperative rehabilitation programs include thermal therapy, electrical therapy, manual therapy, and therapeutic exercise.

SUMMARY:
During the rehabilitation process after rotator cuff repair surgery, patients suffer from increased pain and discomfort due to dysfunction. Pain neuroscience education, a more modern educational method, has been reported to be effective in controlling pain by reducing the fear of movement based on an understanding of neurophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* In case of 4 weeks after receiving arthroscopic rotator cuff repair
* If you wish to participate in research

Exclusion Criteria:

* 65 years old or older
* Those who are limited in conducting education remotely
* If the tear area is large and augmentation is performed
* If there is a previous surgical history at the surgical site
* Osteoarthritis in the shoulder joint
* If you cannot understand the guidelines for evaluation or intervention
* Mental health and cognitive problems

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change in pain intensity from baseline to weeks 2, 4, and 6
  A numeric pain rating scale (NPRS) consisting of 11 points in total from 0 points (no pain) to 10 points (the most severe pain imaginable) is used. The lower the score, the less the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The Better Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes